CLINICAL TRIAL: NCT05029531
Title: Prospective Single Group Study Combined Immuno-hemotherapy for Patients With B-linear Acute Lymphoblastic Leukemia Diagnosed From 0 to 365 Days of Life (ALL-Baby-2021)
Brief Title: Combined Immuno-chemotherapy for Patients With B-linear Acute Lymphoblastic Leukemia Diagnosed From 0 to 365 Days of Life (ALL-Baby-2021)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI-2021-03
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric; ALL, Infants
Keywords: Acute lymphoblastic leukemia; children; infant; treatment сhemotherapy; Immunotherapy; Blinatumomab; Stemm Cell Transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy; Hematopoietic Stem Cell Transplantation; Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention/treatment (Experimental)
  Interventions: Combination Product: the risk-adapted choice of therapy and the use of a combination of chemotherapy with immunotherapy and hematopoietic stem cell transplantation for patients with risk factors.

INTERVENTIONS:
Combination Product: the risk-adapted choice of therapy and the use of a combination of chemotherapy with immunotherapy and hematopoietic stem cell transplantation for patients with risk factors. — two-stage stratification into risk groups: Initially and According to the results of induction therapy MRD-positive patients receive a course of blinatumomab and HSCT.

SUMMARY:
The innovation of this protocol is the risk-adapted choice of therapy and the use of a combination of chemotherapy with immunotherapy and hematopoietic stem cell transplantation for patients with risk factors. Investigators have proposed a two-stage stratification into risk groups:

Initially:

* Standard risk: patients with no rearrangement of the KMT2A gene.
* Intermediate risk: patients with rearrangement of the KMT2A gene without damage to the central nervous system.
* High risk: patients with rearrangement of the KMT2A gene with lesions of the central nervous system.

According to the results of induction therapy:

* The high-risk group includes patients from the standard risk group with an MRD level of more than 0.1% after the induction course and from the intermediate risk group with MRD-positive (PCR) after HR1 block.
* The allocation of children in the first year of life without the rearranged KMT2A gene into a separate group seems to be logical, since the prognosis in this group is better than in children with the rearranged KMT2A gene. In this protocol, non-intensive therapy with consolidations and maintenance therapy remains for those who achieve a low MRD level (less than 0.1%) after a course of induction. The rest of the patients move into a high-risk group: they receive blinatumomab and HSCT.
* The concept of therapy for patients at intermediate risk is based on the rate at which MRD-negativity is achieved: standard consolidation and maintenance therapy for those who became MRD-negative at the end of induction, "block" chemotherapy for those who were positive at the end of induction, but achieved negativity after HR1 block, blinatumomab with HSCT for those who have preserved the MRD after the HR1 block.
* For high-risk patients, a combination of immunotherapy (blinatumomab - a bispecific CD3 / CD19 T-cell activator) and HSCT in the first remission was chosen.

DETAILED DESCRIPTION:
* Standard risk group:
* Induction of remission: 36 days of dexamethasone, 5 weekly injections of vincristine, 2 injections of daunorubicin on days 8 and 22, a single injection of pegelated asparaginase on days 5-7 and 6 weekly intrathecal injections of three drugs (methotrexate, cyamethosar and dexamethason ).
* Further therapy in this therapeutic group depends on the status of remission, the level of MRD on the 36th day of therapy.
* MRD-negative patients receive consolidation therapy in the amount of 3 consolidations (6-mercaptopurine, methotrexate, peg-asparaginase, daunorubicin) with re-induction courses (dexamethasone, vincristine) and maintenance therapy (6-mercaptopurine, methotrexate).
* MRD-positive patients receive a course of blinatumomab and HSCT.
* Intermediate risk group:
* Induction of remission: 36 days of dexamethasone, 5 weekly injections of vincristine, 2 injections of daunorubicin on days 8 and 22, a single injection of pegelated asparaginase on days 5-7, 6 weekly intrathecal injections of three drugs (methotrexate, cyamethosar, dexamethasone).
* Further therapy in this therapeutic group depends on the status of remission on the 36th day of therapy.
* Patients who have achieved molecular remission receive consolidation therapy in the amount of 3 consolidations with re-induction courses and maintenance therapy.
* Patients who have not achieved molecular remission receive HR1 block. Further therapy depends on the remission status after HR1 block. Patients who have not achieved molecular remission receive a course of blinatumomab and HSCT, patients who have achieved molecular remission, two more blocks HR2 and HR3, protocol II and maintenance therapy.
* High risk group:
* Induction of remission: 36 days of dexamethasone, 5 weekly injections of vincristine, 2 injections of daunorubicin on days 8 and 22, a single injection of pegelated asparaginase on days 5-7, 6 weekly intrathecal injections of three drugs (methotrexate, cyamethosar, dexamethasone).
* Further therapy in this therapeutic group does not depend on the status of remission on the 36th day of therapy.
* All patients receive HR1 block, blinatumomab course and HSCT (subject to morphological remission).

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis at 1 to 365 days of life.
* The start of induction therapy within a time interval of study recruitment phase.
* The diagnosis of ALL is to be proved by the morphological, cytochemical, and immunological analysis of tumor cells in bone marrow (see "Diagnostics"). Patients with B-cell (Burkitt) ALL are excluded.
* Informed consent of the patient parents (guardians) to be treated in one of the clinics included in this study.

Exclusion Criteria:

* The disease is a relapse of previously misdiagnosed and, therefore, inadequately treated ALL;
* There is severe concomitant disease, which significantly impedes chemotherapy protocol (such as multiple malformations, heart diseases, metabolic disorders, etc.);
* There is a lack of important data needed for the exact adherence to the cytostatic therapy according to a specific chemotherapy protocol (differential diagnosis of ALL-AML (acute myeloid leukemia) is not possible, stratification according to therapeutic group is not possible);
* The patient was treated before for a long time with cytotoxic drugs;
* There were treatment deviations not covered by the protocol and/or not due to side effects of treatment and/or complications of the disease

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
event free survival | 4 years after the start of therapy
overal survival | 4 years after the start of therapy

SECONDARY OUTCOMES:
risk of relapse | 3 years after the start of therapy
  survival analysis, cumulative risks
frequency of achieving MRD-negative remission | after a course of induction up to 1 week
frequency of achieving MRD-negative remission | after a course of consolidation up to 1 week
mortality associated with HSCT | 2 years post HSCT
  survival analysis, cumulative risks

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology, Moscow, Samory-Mashela,1, Russia

IPD SHARING:
Plan to Share IPD: No